CLINICAL TRIAL: NCT06073860
Title: Reblozyl® (Luspatercept) Post-Marketing Surveillance in Korean Patients With Myelodysplastic Syndrome or Beta Thalassemia
Brief Title: A Post-Marketing Surveillance Study to Assess Safety of Luspatercept in Korean Patients With Myelodysplastic Syndrome or β-thalassemia
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-005
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Myelodysplastic Syndrome; Beta Thalassemia
MeSH Terms: conditions — Myelodysplastic Syndromes; beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with myelodysplastic syndrome or beta thalassemia who will begin luspatercept treatment
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — According to the approved label

SUMMARY:
The purpose of this observational study is to assess the real-world safety of luspatercept in Korean participants with myelodysplastic syndrome (MDS) or beta thalassemia. Investigators will enroll participants who will begin treatment with at least 1 dose of luspatercept.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 19 years of age or older
* Participants who will be treated with luspatercept according to the approved label in the Republic of Korea
* Participants who sign the informed consent form

Exclusion Criteria:

* Participants who are prescribed luspatercept for therapeutic indications not approved in the Republic of Korea
* Participants for whom luspatercept is contraindicated as clarified in the Korean prescribing information approved by the Ministry of Food and Drug Safety

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with transfusion-dependent anemia associated with very low, low, and intermediate-risk myelodysplastic syndrome with ring sideroblasts (MDS-RS) or MDS/myeloproliferative neoplasm with ring sideroblasts and thrombocytosis (MDS/MPN-RS-T) who had an unsatisfactory response to, or are ineligible for erythropoietin-based therapy, and adults with transfusion-dependent anemia associated with beta thalassemia, who will begin therapy with luspatercept.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-12-21 (Estimated); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- South Korea (2):
  - Local Institution - 0001, Seoul
  - Novotech Laboratory Korea Co., Ltd., Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts